CLINICAL TRIAL: NCT04921527
Title: A Multi-center, Double-blind, Randomized Phase III Clinical Trial of Chiauranib Plus Weekly Paclitaxel in Patients with Platinum-refractory or Platinum-resistant Recurrent Ovarian Cancer
Brief Title: Chiauranib Plus Weekly Paclitaxel in Patients with Platinum-refractory or Platinum-resistant Recurrent Ovarian Cancer
Acronym: CHIPRO
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chipscreen Biosciences, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CAR301
Record Dates: First submitted 2021-06-03; First posted 2021-06-10 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Ovarian Cancer; Relapsed or Refractory; Chiauranib; Paclitaxel
MeSH Terms: conditions — Ovarian Neoplasms; Recurrence | interventions — chiauranib; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chiauranib plus weekly paclitaxel (Experimental): Patients receive the combined treatment of chiauranib plus paclitaxel, 21 days for a cycle, 6 cycles at most,Chiauranib is given orally, 50mg once daily. Paclitaxel is given in intravenous infusion on Day 1, 8 and 15. After 6 cycles combined treatment, patients enter the single agent therapy of chiauranib.
  Interventions: Drug: chiauranib; Drug: Paclitaxel
- placebo plus weekly paclitaxel (Placebo Comparator): Patients receive the combined treatment of placebo plus paclitaxel, 21 days for a cycle, 6 cycles at most,placebo is given orally, 50mg once daily. Paclitaxel is given in intravenous infusion on Day 1, 8 and 15. After 6 cycles combined treatment, patients enter the single agent therapy of placebo.
  Interventions: Drug: Placebo; Drug: Paclitaxel

INTERVENTIONS:
Drug: chiauranib — 50mg orally once daily
  Other Names: CS2164
  Arms: Chiauranib plus weekly paclitaxel
Drug: Placebo — 50mg orally once daily
  Arms: placebo plus weekly paclitaxel
Drug: Paclitaxel — at the first cycle, 60mg/m2, i.v infusion on day 1, 8 and 15 ; at the begining of the second cycle, after a comprehensive assessment , investigators decide whether to increase the dosage to 80mg/m2, i.v infusion on day 1, 8 and 15 ;
  Other Names: Anzatax

SUMMARY:
This randomized, double-blind, 2-arm study will evaluate the efficacy and safety of Chiauranib plus weekly paclitaxel versus placebo plus weekly paclitaxel in patients with Platinum-refractory or Platinum-resistant Recurrent ovarian cancer.

DETAILED DESCRIPTION:
Chiauranib is a novel orally active multi-target inhibitor that simultaneously inhibits the angiogenesis-related kinases (VEGFR2, VEGFR1, VEGFR3, PDGFRa and c-Kit), mitosis-related kinase Aurora B and chronic inflammationrelated kinase CSF-1R in a high potency manner with the IC50 at a single-digit nanomolar range. In particular, Chiauranib showed very high selectivity in the kinase inhibition profile with little activity on off-target non-receptor kinases, proteins, GPCR and ion channels, indicative of a better drug safety profile in terms of clinical relevance.

Patients will be randomized to receive treatment with either paclitaxel + Chiauranib or paclitaxel + placebo. Paclitaxel will be repeated every 21 days for a maximum of 6 cycles. Patients with objective response/stable disease after completing 6 courses of chemotherapy will continue Chiauranib or placebo until progression.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to sign a written informed consent document .
* Female, age ≥18 yrs and ≤70 yrs.
* Histological or cytological confirmation of epithelial ovarian cancer, carcinoma tube, or primary peritoneal carcinoma.
* Patients with platinum refractory or platinum resistant ovarian cancer:

  * Platinum refractory: progression during the first platinum-based treatment or within 4 weeks after the first platinum-based primary therapy;
  * Platinum resistant: progression during the platinum-based treatment except for platinum refractory, or within 6 months after the last receipt of platinum-based treatment (patients have received platinum containing chemotherapy at least 4 weeks);
  * Radiological progression during the last treatment administered;
  * no more than 1 prior treatment regimens for recurrent disease.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
* At least 1 lesion can be accurately measured, as defined by RECIST1.1.
* Laboratory criteria are as follows:

  * Complete blood count: hemoglobin (Hb) ≥90g/L ; absolute neutrophil count (ANC) ≥1.5×109/L ; platelets ≥90×109/L;
  * Biochemistry test: serum creatinine(cr) <1.5×ULN; total bilirubin<1.5×ULN; alanine aminotransferase(ALT) ,aspartate aminotransferase(AST)≤2.5×ULN; (ALT,AST≦5×ULN if liver involved) ;
  * Coagulation test: International Normalized Ratio (INR) < 1.5, activeated partial thromboplasting time (APTT) <1.5×ULN
* Life expectancy of at least 3 months.

Exclusion Criteria:

* Patients received vascular endothelial growth factor(VEGF)/vascular endothelial growth factor receptor(VEGFR) inhibitor, like Apatinib, Anlotinib, Fruquintinib, Bevacizumab, etc., or Aurora kinase inhibitors.
* Patients received weekly paclitaxel therapy.
* Has known allegies to Chiauranib, paclitaxel or any of the excipients.
* Biological therapy, immunotherapy, hormonal therapy within 28 days prior to the first dose of study drug.
* prior major surgery or trauma within 14 days prior to first dose of study drug and/or presence of any non-healing wound, fracture, or ulcer.
* Treatment with an investigational agent/instrument within 28 days prior to first dose of study drug.
* Any ongoing toxicity from prior anti-cancer therapy that is >Grade 1.
* Patients with prior invasive malignancies in the past five years with the exception of curatively-treated basal cell or squamous cell carcinoma of the skin or cervical carcinoma in situ.
* History or clinical evidence of central nervous system (CNS) metastases or leptomeningeal carcinomatosis.
* clinically significant central/peripheral nervous system disease.
* Have uncontrolled or significant cardiovascular disease, including:

  * Congestive heart failure, unstable angina pectoris, myocardial infarction within 6 months prior to study entry; arrhythmia, or Left Ventricular Ejection Fraction (LVEF) < 50% requiring treatment with agents during screening stage.
  * primary cardiomyopathy(dilated cardiomyopathy, hypertrophic cardiomyocyte, arrhythmogenic right ventricular cardiomyopathy, restrictive cardiomyopathy, et,al)
  * History of significant QT interval prolongation, or Corrected QT Interval (QTc) > 470 ms prior to study entry
  * Symptomatic coronary heart disease requiring treatment with agents
  * History of hypertension treated by≥2 agents, or the Blood pressure (Bp) ≥140/90 mmHg prior to study entry.
  * Other condition investigator considered inappropriate
* Significant intravenous or arterial thrombosis, such as cerebrovascular accident, pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months.
* History of active bleeding within the past 2 months, patients with bleeding potential during the screening period, or receiving anticoagulation therapy.
* CT or MRI of the chest during the screening period shows interstitial lung disease or pulmonary fibrosis or lung inflammation that requires treatment, or within 6 months before the first dose, history of pneumonia requiring oral or intravenous steroid treatment, history of immune-associated pneumonia after treatment of PD1/PDL1 inhibitor.
* Have clinical significant gastrointestinal abnormality that would impair the ingestion, transportation or absorption of oral agents, history of gastrointestinal perforation or abdominal fistula, peptic ulcer disease within 6 months prior to first dose of study drug or GI obstruction within the past 3 months.
* Pleural fluid, ascites or pericardial effusion with significant symptoms or required treatment of puncture or drainage during the screening period, or history of drainage for therapy within 1 months prior to first dose of study drug.
* Screening for HIV antibody positive.
* Screening test for hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) positive with virus replication, hepatitis C antibody (HCV-Ab) positive with virus replication.
* Active infection requiring oral or intravenous systemic antimicrobial therapy during the screening period.
* Any mental or cognitive disorder, that would impair the ability to understand the informed consent document, or the compliance of study.
* History of organ transplantation or allo-HSCT.
* Any mental or cognitive disorder, that would impair the ability to understand the informed consent document, or the compliance of study.
* Candidates with drug and alcohol abuse.
* Participants of reproductive potential not willing to use adequate contraceptive measures for the duration of the study.Pregnant or breastfeeding women.
* Any other condition which is inappropriate for the study in the opinion of the investigators.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 454 (Estimated)
Dates: Start 2021-12-20 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
progression-free survival (PFS) | assessed up to 1 years
  From the first time of treatment until the date of first documented progression or date of death from any cause, whichever comes first (Assessed by IRC)
overall survival (OS) | assessed up to 2 years
  OS is defined as the length of time from treatment to death from any cause

SECONDARY OUTCOMES:
overall response rate (ORR) | assessed up to 2 years
  ORR is defined as the proportion of participants who have a partial response (PR) or complete response (CR) to therapy according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
duration of response (DOR) | assessed up to 2 years
  From the first date of response until the date of first documented progression
Disease control rate (DCR) | assessed up to 2 years
  DCR is defined as the Proportion of participants in partial, complete or stable desease according to RECIST 1.1. criteria
Quality of life (QoL) | assessed up to 2 years
  QoL assessed by EORTC QLQ-OV28
Toxicity according to NCI CTCAE v5.0 criteria | assessed up to 2 years
  tolerance of the treatment based on AE occurrence according to NCI CTCAE v5.0 criteria
PK parameters of paclitaxel, chiauranib and M345 | assessed up to 2 years
  PK parameters include but not limited to AUC, Cmax, Tmax etc.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohua Wu, Principal Investigator — Fudan university Shanghai cancer centre
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China, China

IPD SHARING:
Plan to Share IPD: No